CLINICAL TRIAL: NCT02336802
Title: The Experimental Study of Threat-Avoidance in Anxiety Patients: Behavioral, Emotional, and Neural Correlates
Brief Title: Threat-Avoidance Learning in Anxiety Patients
Acronym: AVOID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Bram Vervliet, Ph.D., KU Leuven
Other Study IDs: bramvervliet
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Panic Disorder; Phobic Disorders; Stress Disorders, Traumatic
Keywords: Anxiety; Fear; Avoidance
MeSH Terms: conditions — Panic Disorder; Phobic Disorders; Stress Disorders, Traumatic; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy Control Group: Volunteers that meet no diagnostic criteria for mental disorders.
  Interventions: Behavioral: Avoidance experiment
- Panic Disorder Group: Volunteers that meet diagnostic criteria for Panic Disorder.
  Interventions: Behavioral: Avoidance experiment
- Phobic Disorder Group: Volunteers that meet diagnostic criteria for a Phobic Disorder.
  Interventions: Behavioral: Avoidance experiment
- PTSD group: Volunteers that meet diagnostic criteria for Post-Traumatic Stress Disorder
  Interventions: Behavioral: Avoidance experiment

INTERVENTIONS:
Behavioral: Avoidance experiment — Participants complete an avoidance task

SUMMARY:
Anxiety disorders are characterized by exaggerated levels of fear that are not proportional to the actual level of threat. More specifically, anxiety patients have marked deficits in the downregulation of fear reactions during situations of objective safety. Pre-clinical research on Pavlovian fear conditioning and extinction has discovered that fear downregulation stems from areas in the prefrontal cortex (the ventro-medial prefrontal cortex, vmPFC) that recruit intercalated cells in the amygdala to inhibit its central nucleus, which is responsible for a variety of behavioral expressions of fear (Milad & Quirk, 2012). Accordingly, functional magnetic resonance imaging studies (fMRI) revealed reduced vmPFC activity coupled with increased fear reactions during situations of objective safety in anxiety patients (Milad et al., 2009). Another core symptom of anxiety disorders, though much less investigated, is the excessive avoidance of situations that trigger the fears. These 'safety behaviors' often interfere with daily life activities and valued goals in life, and they are thought to perpetuate the exaggerated levels of fear by precluding opportunities to learn that the feared situations are actually not dangerous. Surprisingly, experimental research on avoidance behaviors in anxiety patients is virtually non-existent. This experiment modifies the Pavlovian fear conditioning procedure to include avoidance, and explores the behavioral and neural processes of this type of fear regulation in anxiety patients (trans-diagnostically) and healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age. Proficient in English. Right-handed Free of medication that affect cerebral metabolism. Able to give informed consent. High stress level (defined as a score of >= 3 on the 4-item Perceived Stress Scale).

Exclusion Criteria:

History of neurologic or psychiatric disease (other than the specified anxiety disorder), substance abuse or dependence that is current or within the last year.

Major/chronic medical conditions. History of head injury resulting in prolonged loss of consciousness and/or neurological sequelae. History of seizures. History of stroke Prior neurosurgical procedure. Metal in the body, metal injury to the eyes. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt. Pregnancy; breastfeeding or nursing Claustrophobia Weight > 350 lbs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls, Panic Disorder, Phobic Disorders, Post-Traumatic Stress Disorder
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
functional magnetic resonance imaging | 1.5 hours
  We will measure functional MRI during fear conditioning, avoidance and generalization. Furthermore, we will measure changes in structural MRI data, Diffusion Tensor Imaging (DTI) data and resting state fMRI data.

SECONDARY OUTCOMES:
Skin conductance reactivity | 1.5 hours
  fluctuations in skin conductance will be measured alongside MRI data collection, as a peripheral physiological measure of fear.
Questionnaires | 2 hours
  In a separate sessions, participants will fill out a variety of personality questionnaires probing levels of anxiety and avoidance tendency.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Hermans, Prof., Principal Investigator — University of KU Leuven
Locations (1):
- University of KU Leuven, Leuven, Belgium

REFERENCES:
- [Background] Milad MR, Pitman RK, Ellis CB, Gold AL, Shin LM, Lasko NB, Zeidan MA, Handwerger K, Orr SP, Rauch SL. Neurobiological basis of failure to recall extinction memory in posttraumatic stress disorder. Biol Psychiatry. 2009 Dec 15;66(12):1075-82. doi: 10.1016/j.biopsych.2009.06.026. Epub 2009 Sep 12. PMID 19748076
- [Background] Milad MR, Quirk GJ. Fear extinction as a model for translational neuroscience: ten years of progress. Annu Rev Psychol. 2012;63:129-51. doi: 10.1146/annurev.psych.121208.131631. PMID 22129456